CLINICAL TRIAL: NCT04576507
Title: Effects of Repeated Cannabis Administration on Experimental Pain and Abuse Liability in Humans
Brief Title: Repeated Cannabis Administration on Experimental Pain and Abuse Liability
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Alkermes, Inc. (Industry)
Responsible Party: Principal Investigator, Caroline A. Arout, Ph.D., Assistant Professor of Clinical Neurobiology (in Psychiatry), New York State Psychiatric Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 8016
Record Dates: First submitted 2020-09-29; First posted 2020-10-06 (Actual); Results first posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Cannabis; Pain; Tolerance; Hyperalgesia
MeSH Terms: conditions — Marijuana Abuse; Pain; Hyperalgesia

STUDY DESIGN:
Intervention Model Description: This study comprises a 16-day inpatient stay. On the first full inpatient day (Day 1), participants will smoke one specified strength (Dose A; active cannabis, 2.98% THC and 4.91% CBD) of cannabis. Days 2-8 will comprise Phase 1, in which a second strength (Dose B; placebo cannabis, <0.01% THC,CBD) of cannabis will be administered 3x/day. The next 7 days (Day 9-15) will be Phase 2, in which cannabis Dose A (active cannabis, 2.98% THC and 4.91% CBD) will be administered once again, at the same 3 daily time points.
Masking Description: Participants are blind to what cannabis dose they are receiving on which day, though it is the same for all:
  Day 1: active cannabis (2.98% THC and 4.91% CBD) Day 2-8: placebo cannabis (<0.01% THC, CBD) Day 9-15: active cannabis (2.98% THC and 4.91% CBD)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose A: Standardization Phase (Experimental): On the first full inpatient day (Day 1), participants will smoke one specified strength (Dose A; 75% of active cannabis cigarette, 2.98% THC, 4.91% CBD) of cannabis.
  Interventions: Drug: Active Cannabis
- Dose B: Placebo Phase (Placebo Comparator): Days 2-8 comprises the Placebo phase, in which a second strength (Dose B; 75% of one placebo cannabis cigarette, <0.01% THC, CBD) of cannabis will be administered 3x/day.
  Interventions: Drug: Placebo Cannabis
- Dose A: Active Phase (Experimental): Days 9-15 comprise the Active Phase, cannabis Dose A (75% of one active cannabis cigarette, 2.98% THC, 4.91% CBD) will be administered once again, 3x/day.
  Interventions: Drug: Active Cannabis

INTERVENTIONS:
Drug: Active Cannabis — 2.98% THC:4.91% CBD cannabis.
  Arms: Dose A: Active Phase; Dose A: Standardization Phase
Drug: Placebo Cannabis — <0.01% THC:CBD cannabis.
  Arms: Dose B: Placebo Phase

SUMMARY:
Chronic pain is a significant public health concern in the U.S., for which prescription opioids have historically been the standard treatment. This has resulted in striking rates of opioid use disorders and fatal overdoses. Identifying non-opioid medications for the management of chronic pain with minimal abuse liability is a public health necessity, and cannabinoids are a promising drug class for this purpose. More than 80% of medicinal cannabis users report pain as their primary medical indication. These patients tend to seek products that are low in delta-9-tetrahydrocannabinol (THC; the primary psychoactive, and thus intoxicating, component of cannabis), and high in cannabidiol (CBD), a cannabinoid that purportedly has therapeutic benefit for pain but does not produce intoxicating effects. However, there are few well-controlled human laboratory studies assessing the efficacy of high-CBD cannabis for pain in the context of abuse, and even less is known regarding the effects of daily repeated use of cannabis on pain and its relationship to abuse liability.

The proposed randomized, within-subjects, placebo-controlled 16-day crossover inpatient human laboratory pilot study (N = 16 healthy cannabis users; 8 men, 8 women) will address important gaps in our understanding of the potential therapeutic utility of cannabis for pain: 1) If repeated cannabis use can result in hyperalgesia; 2) If tolerance to the analgesic and abuse-related effects of cannabis develops and is reversible. Two distinct modalities of experimental pain will be assessed: The Cold Pressor Test (CPT) and Quantitative Sensory Testing Thermal Temporal Summation (QST-TTS), and participants will smoke cannabis 3x/day. Throughout the study, experimental pain and abuse-related effects will be assessed, as will sleep and subjective mood assessments.

This protocol is currently suspended due to the NYSPI human subjects research pause and results cannot currently be analyzed and posted. Upon un-suspension, we will analyze the data and post results immediately.

ELIGIBILITY:
Inclusion Criteria:

* Males/non-pregnant females, 21-60 years old
* Current cannabis user
* Able to perform all study procedures

Exclusion Criteria:

* Use of other illicit drugs
* If medical history, physical and psychiatric examination, or laboratory tests performed during the screening process reveal any significant illness that the study physician deems contraindicated for study participation
* Insensitivity to the cold-water stimulus of the Cold Pressor Test or the heat stimulus of Quantitative Sensory Testing

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between June 2021 and June 2023. Eligible participants were recruited from the New York, NY area and occurred through advertisements in local newspapers, online through Craigslist, RecruitMe, and by word of mouth.
Pre-assignment Details: There were no significant events in the study post-enrollment and/or prior to participants beginning study procedures.
Groups:
- Dose A - Dose B - Dose A: On the first full inpatient day (Day 1), participants smoked one specified strength (Dose A; active cannabis, 2.98% THC, 4.91% CBD) of cannabis. Days 2-8 comprised Phase 1, in which a second strength (Dose B; placebo cannabis, <0.01% THC, CBD) of cannabis was administered 3x/day. The next 7 days (Day 9-15) comprised Phase 2, in which cannabis Dose A (active cannabis, 2.98% THC, 4.91% CBD) was administered again, at the same 3 daily time points. All participants underwent this same allocation.
  Cannabis: Investigates two strengths of cannabis.
Period: Overall Study
Arm/Group | Dose A - Dose B - Dose A
Started | 10
Completed (Of the 10 that were enrolled and started the study, five did not complete the entire study (4 because of an Adverse Event; 1 because they chose not to continue).) | 5
Not Completed | 5
Not completed — Adverse Event | 4
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Dose A - Dose B - Dose A
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 0
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Cold Pressor Test (CPT) Latency
Description: The CPT apparatus consists of two refrigerated circulators, filled with warm (36.5-37.5°C). participants will complete the CPT 30 minutes before the 1000h cannabis administration (baseline), and 15, 30, 45, 60, and 90 minutes post-cannabis administration. and cold (3.5 - 4.5°C) water. Participants will insert their non-dominant hand into the warm water and remove it after 3 minutes; skin temperature of the thumb pad will be measured. Participants will then insert their hand in the cold water and will be instructed to report when they first experience pain (pain threshold) and remove their hand when the cold water can no longer be tolerated (pain tolerance). Maximum immersion time will be 3 minutes.
  Data points reported here represent Percent Change in Pain Tolerance from Day 1 (first timepoint, 15 minutes post-cannabis [2.98% THC / 4.91% CBD]) across study days (Day 2, 5, 8, 9, 12, and 15). Other timepoints are not reported.
Time Frame: Up to 15 days
Population: Data represents CPT Pain Tolerance for study completers (n=5) across the 15-day testing period. This is a repeated measures design, meaning that all 5 participants contributed to each timepoint.
Measure: Mean (Standard Error); unit: percent change from Day 1 baseline
Groups:
- CPT Pain Tolerance: Day 2; CPT Pain Tolerance: Day 5; CPT Pain Tolerance: Day 8; CPT Pain Tolerance: Day 9; CPT Pain Tolerance: Day 12; CPT Pain Tolerance: Day 15: The CPT apparatus consists of two refrigerated circulators, filled with warm (36.5-37.5°C). participants will complete the CPT 30 minutes before the 1000h cannabis administration (baseline), and 0, 15, 30, 45, 60, and 90 minutes post-cannabis administration. and cold (3.5 - 4.5°C) water. Participants will insert their non-dominant hand into the warm water and remove it after 3 minutes; skin temperature of the thumb pad will be measured. Participants will then insert their hand in the cold water and will be instructed to report when they first experience pain (pain threshold) and remove their hand when the cold water can no longer be tolerated (pain tolerance). Maximum immersion time will be 3 minutes.
  Data points represent Percent Change in Pain Tolerance from Day 1 (first timepoint, 15 minutes post-cannabis [2.98% THC / 4.91% CBD]) across study days (Day 2, 5, 8, 9, 12, and 15).
Arm/Group | CPT Pain Tolerance: Day 2 | CPT Pain Tolerance: Day 5 | CPT Pain Tolerance: Day 8 | CPT Pain Tolerance: Day 9 | CPT Pain Tolerance: Day 12 | CPT Pain Tolerance: Day 15
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5
percent change from Day 1 baseline | 21.40 (24.22) | 10.94 (18.81) | 2.07 (5.84) | 15.17 (16.97) | 20.06 (25.07) | 30.16 (28.67)

2. Secondary Outcome: Change in Cannabis Rating Form (CRF) Ratings
Description: Participants rate the "high" experienced as a result of cannabis administration on a 100mm visual analog scale. Data points represent Percent Change from Day 1 (first timepoint, 15 minutes post-cannabis [2.98% THC / 4.91% CBD]) across study days (Day 2, 5, 8, 9, 12, and 15)
  Repeats at days 1, 2, 5, 8, 9, 12, and 15.
Time Frame: Up to 15 days
Population: Data represents mean ratings for "high" on a 0-100mm visual analog scale, where 0 represents no "high" and 100 represents the maximum amount of "high" for study completers (n=5) across the 15-day testing period. This is a repeated measures design, meaning that all 5 participants contributed to each timepoint.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Day 1 Cannabis Rating Form: "High"; Day 2 Cannabis Rating Form: "High"; Day 5 Cannabis Rating Form: "High"; Day 8 Cannabis Rating Form: "High"; Day 9 Cannabis Rating Form: "High"; Day 12 Cannabis Rating Form: "High"; Day 15 Cannabis Rating Form: "High": Participants rate the "high" experienced as a result of cannabis administration on a 100mm visual analog scale. Data points represent Percent Change from Day 1 (first timepoint, 15 minutes post-cannabis [2.98% THC / 4.91% CBD]) across study days (Day 2, 5, 8, 9, 12, and 15) Repeats at days 1, 2, 5, 8, 9, 12, and 15.
Arm/Group | Day 1 Cannabis Rating Form: "High" | Day 2 Cannabis Rating Form: "High" | Day 5 Cannabis Rating Form: "High" | Day 8 Cannabis Rating Form: "High" | Day 9 Cannabis Rating Form: "High" | Day 12 Cannabis Rating Form: "High" | Day 15 Cannabis Rating Form: "High"
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5 | 5
score on a scale | 14.60 (7.53) | 9.6 (7.756) | 17.60 (12.66) | 11.20 (8.16) | 30.80 (10.29) | 42.00 (18.20) | 41.40 (15.84)

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected continuously for the duration of study participation for each participant, which was approximately 1 month (screening through study completion). All participants received the same order of drug administration and as such, are reported under one condition.
Description: Drug effects as a result of cannabis administration were expected, and not considered adverse events at the time.
Groups:
- All Participants: Data on potential adverse events were collected throughout the duration of the study (06/2021 - 06/2023).
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 4/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=10)
High blood pressure (Cardiac disorders) | 1 (1) — Pre-active cannabis (before Dose A)
Acid reflux (Gastrointestinal disorders) | 1 (1) — During placebo cannabis administration (Dose B).
High blood pressure (Cardiac disorders) | 1 (1) — During active cannabis administration (Dose A)
High blood pressure (Cardiac disorders) | 1 (1) — During placebo cannabis administration (Dose B).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2025-02-10): https://cdn.clinicaltrials.gov/large-docs/07/NCT04576507/Prot_000.pdf
  • Statistical Analysis Plan (2025-04-14): https://cdn.clinicaltrials.gov/large-docs/07/NCT04576507/SAP_001.pdf